CLINICAL TRIAL: NCT02214108
Title: Effect of Physical Activity Trough Interactive Video Games in Overweight, Randomized, Controlled Study.
Brief Title: Effect of Physical Activity Through Interactive Video Games in Overweight Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Giuseppe Grandy, Medical head of Nutrition Center Albina Patino, Centro Pediatrico Albina de Patino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: protwii2013
Record Dates: First submitted 2014-07-25; First posted 2014-08-12 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Overweight
Keywords: BMI; Obesity; overweight; child; Physical activity
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phisical activity with Nintendo Wii (Experimental): 3 hours of weekly of physical activity, divided in 1 hour interday with Nintendo WII. games applied: Wii Boxing, Wii Tennis; Wii Bowling
  Interventions: Other: Nintendo Wii
- phisical activity with phisiotherapist (No Intervention): 3 hours of weekly physical activity, divided in 1 hour interday. applying cardiovascular and muscular endurance static exercises.

INTERVENTIONS:
Other: Nintendo Wii — Tennis, box and bowling on Nintendo Wii, 3 hours per week.
  Other Names: active video games
  Arms: Phisical activity with Nintendo Wii

SUMMARY:
The purpose of this study is to determine the effect of interactive video game in management of overweight in children. The investigators will evaluate the effect of product versus standard physical activity.

DETAILED DESCRIPTION:
Background. Child Overweight and obesity are a world public health problem, in low income countries is more. One difficulty in the management is the poor adherence to physical activity, some studies show that active video games could improve this.

Objective: Establish the effect of the introduction of active video game (Nintendo Wii) on fitness, anthropometry and adherence to treatment, as part of an intervention program for the management of childhood obesity in children over 5 years of age with obesity Methodology: A clinical trial, randomized and controlled. children between 5-10 years with a diagnosis of overweight or obese, were divided into two groups. (Wii group), received 3 weekly sessions of one hour of physical activity by an active video game, the other group (control group) received 3 weekly sessions of one hour of physical activity by static exercises.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5-10 years with a diagnosis of overweight or obese (according to WHO criteria)

Exclusion Criteria:

* overweight or obese due other disease.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | one month

SECONDARY OUTCOMES:
change in weight | one month
change in physical endurance | one month
variations in serum lipids | 1 month
  Cholesterol, triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Esteban Grandy Aranda, MSc, Study Director — Centro de Pediatria Albina Patino; Alicia Ribero Nogales, MD, Principal Investigator — Centro de Pediatria Albina Patino; Gerardo Weisstaub, MSc, Study Chair — Institute of Nutrition and Technology of Food.
Locations (1):
- Pediatric Center Albina Patino, Cochabamba, Departamento de Cochabamba, Bolivia